CLINICAL TRIAL: NCT05910801
Title: Tafasitamab, Lenalidomide and Venetoclax Combination Therapy for Relapsed or Refractory Mantle Cell Lymphoma (V-MIND): a Phase II Study with Safety Lead-In
Brief Title: Tafasitamab, Lenalidomide and Venetoclax for the Treatment of Relapsed or Refractory Mantle Cell Lymphoma
Acronym: V-MIND
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Academic and Community Cancer Research United (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACCRU-LY-2101; NCI-2023-03968 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ACCRU-LY-2101 (Other: Academic and Community Cancer Research United); P30CA015083 (NIH)
Record Dates: First submitted 2023-06-09; First posted 2023-06-20 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Recurrent Mantle Cell Lymphoma; Refractory Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — Biopsy; Specimen Handling; Lenalidomide; Spinal Puncture; Magnetic Resonance Spectroscopy; tafasitamab; Immunoglobulins; Disulfides; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Tafasitamab, lenalidomide, venetoclax) (Experimental): Patients receive tafasitamab IV, lenalidomide PO and venetoclax PO while on study. Patients may undergo lumbar puncture during screening. Patients undergo CT scan and blood sample collection and may undergo MRI and tumor biopsy on study and during follow-up. Patients undergo PET/CT, bone marrow biopsy, and bone marrow aspirate throughout the study.
  Interventions: Procedure: Biopsy; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Drug: Lenalidomide; Procedure: Lumbar Puncture; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Biological: Tafasitamab; Drug: Venetoclax

INTERVENTIONS:
Procedure: Biopsy — Undergo biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT Scan; tomography
Drug: Lenalidomide — Given PO
  Other Names: CC-5013; CC5013; CDC 501; Revlimid
Procedure: Lumbar Puncture — Undergo lumbar puncture
  Other Names: LP; Spinal Tap
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Procedure: Positron Emission Tomography — Undergo PET/CT scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
Biological: Tafasitamab — Given IV
  Other Names: Immunoglobulin, Anti-(Human Cd19 Antigen) (Human-mus musculus Monoclonal MOR00208 Heavy Chain), Disulfide with Human-mus musculus Monoclonal MOR00208 .Kappa.-chain, Dimer; Monjuvi; MOR-00208; MOR00208; MOR208; Tafasitamab-cxix; XmAb5574
Drug: Venetoclax — Given PO
  Other Names: ABT-0199; ABT-199; ABT199; GDC-0199; RG7601; Venclexta; Venclyxto

SUMMARY:
This phase II trial tests how well tafasitamab, lenalidomide and venetoclax work in treating patients with mantle cell lymphoma that has come back (after a period of improvement) (relapsed) or that has not responded to previous treatment (refractory). Tafasitamab is a monoclonal antibody that may interfere with the ability of cancer cells to grow and spread. Lenalidomide is in a class of medications called immunomodulatory agents. It works by helping the immune system kill cancer cells. Venetoclax is in a class of medications called B-cell lymphoma-2 (Bcl-2) inhibitors. It may stop the growth of cancer cells by blocking Bcl-2, a protein needed for cancer cell survival. Giving tafasitamab, lenalidomide and venetoclax together may kill cancer cells more efficiently in patients with relapsed or refractory mantle cell lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the overall response rate in patients with relapsed/refractory mantle cell lymphoma after treatment with tafasitamab, lenalidomide and venetoclax combination.

SECONDARY OBJECTIVES:

I. To estimate the complete response rate in patients with relapsed/refractory mantle cell lymphoma after treatment with tafasitamab, lenalidomide and venetoclax combination.

II. To estimate the duration of response (DoR) in patients with relapsed/refractory mantle cell lymphoma after treatment with tafasitamab, lenalidomide and venetoclax combination.

III. To estimate the progression free survival (PFS) in patients with relapsed/refractory mantle cell lymphoma after treatment with tafasitamab, lenalidomide and venetoclax combination.

IV. To estimate the overall survival (OS) in patients with relapsed/refractory mantle cell lymphoma after treatment with tafasitamab, lenalidomide and venetoclax combination.

V. To evaluate the safety profile of tafasitamab, lenalidomide and venetoclax combination in patients with relapsed/refractory mantle cell lymphoma.

CORRELATIVE OBJECTIVES:

I. To assess the rate of undetectable minimal residual disease (uMRD) in peripheral blood by multi-color flow cytometry.

II. To assess the correlation between MRD status with clinical outcomes such as DoR, PFS and OS.

OUTLINE: Patients receive tafasitamab intravenously (IV), lenalidomide orally (PO) and venetoclax PO while on study. Patients may undergo lumbar puncture during screening. Patients undergo computed tomography (CT) scan and blood sample collection and may undergo magnetic resonance imaging (MRI) and tumor biopsy on study and during follow-up. Patients undergo positron emission tomography (PET)/CT, bone marrow biopsy, and bone marrow aspirate throughout the study.

After treatment completion, patients follow up every 3 months for 1 year, every 4 months for 1 year and then every 6 months until up to 5 years after entering the trial.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years old
* Confirmed pathology diagnosis of mantle cell lymphoma (MCL) with t(11;14)(q13;q32) translocation or cyclin D1 overexpression NOTE: Patients with relapsed/refractory MCL after prior anti-CD19 therapy (such as chimeric antigen receptor [CAR] T-cell therapy) should have confirmed preserved expression of CD19, unless a biopsy is not feasible or associated with a high risk of complications in the treating physician's opinion
* Relapsed or refractory disease, which is defined as patients with >= 1 line of prior systemic treatment NOTE: Prior exposure to lenalidomide or venetoclax is allowed, provided there was no disease progression on lenalidomide or venetoclax
* In the view of the treating physician, the patient is in need of treatment, for example, with lymphoma-related symptoms or cytopenia
* Evaluable disease, which is defined as at least one lymph node or other type of lesion that has a size >= 1.5 cm, or spleen size >= 15 cm or white blood cell (WBC) >= 30,000/mm^3 in leukemic non-nodal MCL patients
* Eastern Cooperative Oncology Group Performance Status (PS) 0, 1, or 2
* Absolute neutrophil count (ANC) >= 1500/mm^3 (obtained =< 14 days prior to registration)
* Platelet count >= 75,000/mm^3 (>= 50,000/mm^3 if there is evidence of bone marrow involvement by MCL or hypersplenism) (obtained =< 14 days prior to registration)
* Hemoglobin > 8.0 g/dL (obtained =< 14 days prior to registration)
* Activated partial thromboplastin time (aPTT) or partial thromboplastin time (PTT) =< 1.5 × upper normal limit (ULN) (obtained =< 14 days prior to registration)
* Prothrombin (PT) or international normalized ratio (INR) =< 1.5 × upper normal limit (ULN) (obtained =< 14 days prior to registration)
* Total bilirubin =< 1.5 × ULN (or =< 3 × ULN if there is evidence of parenchymal liver involvement with MCL or documented Gilbert's disease) (obtained =< 14 days prior to registration)
* Alanine aminotransferase (ALT) and aspartate transaminase (AST) =< 3 × ULN (or =< 5 × ULN if there is evidence of parenchymal liver involvement with MCL) (obtained =< 14 days prior to registration)
* Calculated creatinine clearance > 60 ml/min using the Cockcroft-Gault formula (obtained =< 14 days prior to registration)
* Negative pregnancy test done =< 7 days prior to registration, for women of reproductive potential only NOTE: If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required NOTE: Females of reproductive potential include all females who are menstruating, amenorrheic from previous medical treatments, under 50 years of age, and/or perimenopausal, and do not qualify for the females not of reproductive potential category. Females not of reproductive potential include females who have been in natural menopause for at least 24 consecutive months, or who have had a hysterectomy and/or bilateral oophorectomy, or female children who have not started menstruating
* Agree to use effective contraception during study treatment and for 4 weeks after last dose of lenalidomide and for 3 months after last dose of tafasitamab (whichever is longer) Females of reproductive potential must commit either to abstain continuously from heterosexual sexual intercourse or to use two methods of reliable birth control simultaneously: one highly effective form of contraception - tubal ligation, intrauterine device (IUD), hormonal (birth control pills, injections, hormonal patches, vaginal rings, or implants), or partner's vasectomy, and one additional effective contraceptive method - male latex or synthetic condom, diaphragm, or cervical cap. Contraception should continue during therapy, during dose interruptions, and for 4 weeks following discontinuation of lenalidomide and for 3 months after discontinuation of tafasitamab (whichever is longer). Reliable contraception is indicated even where there has been a history of infertility, unless due to hysterectomy. If needed, females of reproductive potential should be referred to a qualified provider of contraceptive methods Males must always use a latex or synthetic condom during any sexual contact with females of reproductive potential during trial therapy, during dose interruptions, and for 4 weeks following discontinuation of lenalidomide and for 3 months after discontinuation of tafasitamab (whichever is longer), even if they have undergone a successful vasectomy. Male patients must not donate sperm
* Willing to be registered into the mandatory REVLIMID REMS (trademark) program, and willing and able to comply with the requirements of the REVLIMID REMS program
* Able to take low-dose aspirin (81 mg) daily or an alternative form of anticoagulation
* Subject must voluntarily sign and date an informed consent =< 28 days prior to registration
* Willing to return to enrolling institution for follow-up during the active monitoring phase (i.e., active treatment and clinical follow-up) of the study
* Willing to provide mandatory blood specimens for correlative research and banking for future correlative research pertinent to this study

Exclusion Criteria:

* Any of the following:

  * Pregnant persons
  * Nursing persons (lactating persons are eligible provided that they agree not to use their breast milk to feed while receiving treatment on the study or within 3 months of the last dose of study treatment)
  * Men or women of reproductive potential who are unwilling to employ adequate contraception during treatment and for 4 weeks after last dose of lenalidomide or for 3 months after last dose of tafasitamab (whichever is longer)
* Any of the following prior therapies:

  * Autologous stem cell transplant =< 90 days prior to registration
  * Allogeneic stem cell transplant
  * Anti-CD19 CAR T-cell therapy =< 90 days prior to registration
* Any central nervous system (CNS) involvement by MCL (e.g., any parenchymal, leptomeningeal, cerebrospinal fluid [CSF], cranial or spinal nerve root involvement)
* Receiving any other treatment which would be considered as a treatment for MCL (with the exception of corticosteroid). If a patient received recent MCL treatment prior to registration, at least 5 half-lives of the drug(s) OR 14 days must have passed following the last dose for the patient to be eligible
* Any of the following medication requirement or recent use:

  * Anticoagulation with a vitamin K antagonist =< 7 days prior to registration
  * Requirement of a P-gp inhibitor during the study
  * Requirement of a strong cytochrome P450 (CYP) 3A inhibitor or inducer during the study
  * Use of a strong or moderate CYP3A inhibitor or inducer =< 7 days prior to registration

NOTE: Because of their effect on CYP3A4, use of any of the following within 3 days of registration or planned use during study participation is prohibited:

* Grapefruit or grapefruit products
* Seville oranges or products from Seville oranges
* Star fruit

  * Human Immunodeficiency Virus (HIV) positive. All subjects will be screened for HIV =< 14 days prior to registration
  * Patient with chronic hepatitis B virus (HBV) or hepatitis C (HCV) requiring treatment. All subjects will be screened for hepatitis B and hepatitis C =< 14 days prior to registration NOTE: Patients with positive hepatitis B surface antigen (HBsAg) are excluded from participation in this trial. Patients with positive hepatitis B core antibody (anti-HBc) and negative HBsAg require hepatitis B polymerase chain reaction (PCR) evaluation. Patients who are hepatitis B PCR positive will be excluded from participating in this trial NOTE: Patients with positive hepatitis C antibody need to have a negative result for hepatitis C ribonucleic acid (RNA). Patients who are hepatitis C RNA positive will be excluded from participating in this trial
  * Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the local investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
  * Uncontrolled intercurrent illness, in the judgement of the local investigator, including, but not limited to:
* New York Heart Association (NYHA) class III or IV or symptomatic congestive heart failure
* Unstable angina or acute coronary syndrome =< 3 months prior to registration
* Uncontrolled or symptomatic cardiac arrhythmia

  * NOTE: Patients with pacemakers are eligible if they have no history of fainting or clinically relevant arrhythmias while using the pacemaker
* Oxygen dependent baseline lung disease (such as interstitial lung disease or chronic obstructive pulmonary disease [COPD])
* Ongoing inflammatory bowel disease (such as ulcerative colitis) requiring active treatment
* Ongoing malabsorption syndrome or other condition that precludes enteral route of administration
* Ongoing or active infection (viral, bacterial, or fungal)
* Psychiatric illness/social situations that would limit compliance with study requirements

  * History of the following:
* Cerebral vascular accident within 24 weeks prior to registration
* Myocardial infarction within 24 weeks prior to registration
* Major surgery =< 28 days prior to registration
* Live vaccination =< 28 days prior to registration
* Life-threatening thrombosis/embolism
* Bleeding diathesis that precludes the use of low-dose aspirin (81 mg daily) or any form of anticoagulation

  * Other active primary malignancy (other than localized non-melanotic skin cancer or carcinoma in situ of the cervix) requiring treatment or limiting expected survival to =< 2 years NOTE: If there is a history of prior malignancy, the patient must be in remission not require ongoing therapy such as radiation, chemotherapy or immunotherapy for their cancer. Patients on adjuvant hormonal therapy for adequately treated nonmetastatic breast or prostate cancer are permitted if they meet other eligibility criteria
  * Unable to swallow oral drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-01-04 (Actual); Primary Completion 2029-12-30 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | Up to 5 years
  A response is defined to be either a partial metabolic response (PMR) or complete metabolic response (CMR) by positron emission tomography (PET) or a partial response (PR) or complete response (CR) by computed tomography (CT) noted as the objective status using Lugano criteria. Objective response rate is defined as the proportion of evaluable patients who achieve response while on treatment. Estimate and corresponding 95% confidence intervals will be calculated according to the approach of Duffy and Santner.

SECONDARY OUTCOMES:
Complete response rate | Up to 5 years
  Will be estimated for each cohort by the total number of patients who achieve a CMR (by PET/CT) or CR (by CT) at any time on treatment divided by the total number of evaluable patients. Point estimate for complete response rate and corresponding 95% confidence interval will be provided using exact method.
Duration of response | From first documentation of objective status(PMR or CMR by PET/CT, or PR or CR by CT) to the earliest date of progression or death, assessed up to 5 years
  Will be estimated using the method of Kaplan-Meier separately for each cohort.
Progression free survival | From registration to the earliest date of documentation of disease progression or death due to any cause, assessed up to 5 years
  Will be estimated using method of Kaplan-Meier separately for each cohort.
Overall survival | From registration to death due to any cause, assessed up to 5 years
  Will be estimated using method of Kaplan-Meier for each cohort.
Incidence of adverse events (AE) | Up to 5 years
  The maximum grade for each type of AE from each patient will be used for analysis, and frequency tables will be reviewed to determine patterns. Additionally, the relationship of the AE(s) to the study treatment will be taken into consideration. Adverse events will be reported separately for each cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Yucai Wang, Principal Investigator — Academic and Community Cancer Research United
Locations (2):
- United States (2):
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - M D Anderson Cancer Center, Houston, Texas